CLINICAL TRIAL: NCT05421481
Title: The Effect Of Multiple Nursing Interventions Of Physical Activity And on Health Promotion In The Elderly: Randomized Controlled Experiment
Brief Title: Elderly Health Promotion and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Sacikara, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22149001
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Behavior, Health
Keywords: health promotion; physical activity; health promotion model; mobile application
MeSH Terms: conditions — Health Behavior; Motor Activity | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In the first interview, the mobile phone contact information of the elderly will be obtained and planning will be made for the first home visit when appropriate. Physical activity education and health promotion during home visit brochure will be provided. A brochure containing healthy lifestyle habits, health responsibility, exercise, nutrition, oral hygiene and social support behaviors will be provided for general health promotion awareness. The Google Fit application, which is a mobile application, will be downloaded to the phones of the people and installed together, how to use the application will be explained and the application will be made. The group walk to be done. A reminder message will be sent by phone. Message content "For your health, you should exercise at least 30 minutes a week for a total of 150 minutes." will be. Groups of five will be formed for the group walking, and it will be completed within seven days.
  Interventions: Other: home visit, health education, mobile application, group walk, message
- control group (No Intervention): There is no health-related practice in the pensioners' club. No intervention will be made in the control group. After the experimental group's attempts are completed, a home visit is planned for the control group, and it is planned to make physical activity training, brochure, google fit application installation attempts.

INTERVENTIONS:
Other: home visit, health education, mobile application, group walk, message — Home visit: Elderly individuals will be visited once at home. During the home visit, training will be given on the slide about physical activity. A brochure will be provided for general health promotion awareness. Counseling will also be provided during the home visit process.
  Google Fit Application: During the home visit, the application will be downloaded to the phone of the elderly, and a document will be given about the use of the application after the usage is explained. The researcher will support those who have problems with the application in the following weeks.
  Group walking: The walk, which will be done once, will be done in a light paced manner, and the purpose of the walk is to see the number of steps in the mobile application and to increase their motivation with the group.
  Message: Message content "For your health, you should exercise at least 30 minutes a week for a total of 150 minutes." will be.
  Arms: intervention group

SUMMARY:
Nurses have an important place in establishing health promotion practices and policies for the elderly to help older adults manage their lifestyles. For health promotion programs to produce reliable results, health promotion programs that will improve public health must be model/theory-based. In line with all these data, although technology applications have been used more and more in recent years, studies with a high level of evidence on the effects of multi-intervention on physical activity and health improvement in the elderly are insufficient. This study will be examined the effects of home visit education, mobile application (Google Fit), group walking, and phone reminder attempts for the elderly between the ages of 60-70, based on Pender's Health Promotion Model, on physical activity and health promotion after 6 months of follow-up.

DETAILED DESCRIPTION:
The proportion of the elderly population is gradually increasing worldwide and in our country. Along with the increasing elderly population, many health problems are also developing and it is seen that the diagnosis and treatment processes cause high financial expenditures. Prevention of chronic diseases, which can reduce the quality of life and independence of elderly individuals and become an important burden for health systems, has become a necessity. Almost all of the chronic diseases are caused by a negative lifestyle and inadequate health promotion efforts. Similar common diseases and causes of death in our country and in the world are mostly cardiovascular diseases, cancer, diabetes and infectious diseases. The modifiable causes of these diseases are also similar. These are tobacco use, nutritional deficiencies, stress and lack of physical activity. Positive health behaviors (nutrition, physical activity, not smoking, stress management) to be gained to individuals can reduce the incidence of these diseases. For this reason, health promotion programs have an important place in bringing positive health behaviors to the individual, family and society. One of the best ways to improve the health of the elderly is physical activity. WHO recommends regular physical activity for all older adults, 3 or more days a week of moderate or higher-intensity variety of multi-component physical activity. A minimal exercise supervision through weekly visits and/or phone calls is recommended to improve the effects of home-based exercise. The use of a pedometer has been shown to significantly increase physical activity in the elderly when a step goal is set. Another piece of evidence has been found that group-based interventions promote the maintenance of targeted behaviors through peer support. Digital behavior change interventions related to physical activity in the elderly (activity meters, pedometer, use of mobile applications, smart wristbands, smart watches) show that they are beneficial for monitoring and promoting physical activity and improving the health of the elderly. Thanks to mobile applications such as Google Fit, health data such as physical activity can be easily tracked, monitored and recorded. It is important to adopt a health promotion approach that allows older individuals to increase their control over their health and accepts healthy aging as a part of aging. In the Eleventh Development Plan of our country, it is aimed to increase the quality of life of the elderly population by creating an environment where the elderly can live independently, actively and healthily in line with their own preferences, and take part in economic and social life. Nurses have an important place in establishing health promotion practices and policies for the elderly to help older adults manage their lifestyles. In order for health promotion programs to produce reliable results, it is very important that health promotion programs that will improve public health are model/theory-based. In line with all these data, although technology applications have been used more and more in recent years, studies with a high level of evidence on the effects of multi-intervention on physical activity and health improvement in the elderly are insufficient. In this study, the effects of home visit education, mobile application (Google Fit), group walk, phone reminder attempts for the elderly between the ages of 60-70, based on Pender's Health Promotion Model, on physical activity and health promotion after 6 months of follow-up. will be examinedIn line with all these data, although technology applications have been used more and more in recent years, studies with a high level of evidence on the effects of multi-intervention on physical activity and health improvement in the elderly are insufficient. In this study, the effects of home visit education, mobile application (Google Fit), group walk, and phone reminder attempts for the elderly between the ages of 60-70, based on Pender's Health Promotion Model, on physical activity and health promotion after 6 months of follow-up will be reviewed.

Method: The project was planned in a pretest-posttest randomized controlled experimental type. The study will be carried out in Melikşah, Havzan and Konevi Pensioners' Club in Meram district of Konya between June 2022 and December 2022. In determining the sample size, based on the study in the literature, the number of samples was determined as 66 in the experimental and control groups, 33 in each group, taking into account the 95% power level and possible losses (20% drop out). Information Form, Elderly Health Promotion Scale, and Elderly Physical Fitness and Exercise Activity Scale will be used to collect study data. Subjects meeting the inclusion criteria who gave informed consent will be randomly assigned to groups using the block randomization technique.

Management: At the beginning of the study, the Information Form, the Elderly Health Promotion Scale and the Physical Fitness and Exercise Activity Scale of the Elderly Individuals, which were the pre-test data, will be collected face to face by the assistant researcher from the elderly individuals aged 60-70 who came to Melikşah, Havzan and Konevi Retirement Club, paying attention to the pandemic conditions; At the end of the 6th month, an independent researcher will fill in the Elderly Health Promotion Scale and the Elderly Physical Fitness and Exercise Activity Scale.

Application:

* Pre-tests of the Information Form, Elderly Health Promotion Scale and the Physical Fitness and Exercise Activity Scale of Elderly Individuals will be applied by obtaining the informed consent of the elderly people who gave their consent to participate in the study. The elderly who consented to participate will be assigned to either the experimental or control group according to the block randomization list previously prepared by an independent statistician.
* At the first meeting, mobile phone contact information of the elderly will be obtained and planning will be made for the first home visit at a time when the elderly are suitable. Physical activity training will be provided during the home visit. A brochure including healthy lifestyle habits, health responsibility, exercise, nutrition, oral hygiene and social support behaviors will be provided for general health promotion awareness. The Google Fit application, which is a mobile application, will be downloaded to the phones of the people and installed together, and how to use the application will be explained and the application will be made. The visit will take a maximum of 40 minutes. A visit was planned for six elderly people in one day and home visits were planned to be completed in a total of six days for the entire experimental group. The data (step count and physical activity duration) of the day before the 2nd week, 10th week and 6th month of the attempt will be recorded from the Google Fit application.
* A reminder message will be sent by phone. From the 2nd week of the initiatives, a message will be sent every Monday at 10:00. Message content "For your health, you should exercise at least 30 minutes a week for a total of 150 minutes." will be.
* Group Walking: Groups of five people will be formed for the group walking (as the number of people to be included in the experimental group is 33, one of the group will be three people) and it will be completed in seven days. The walking will be done in a light paced manner and the purpose of the walking is to see the number of steps in the mobile application and to increase their motivation with the group. People will be invited to the Melikşah park for the group walking. They will be reminded to bring their phones with them.
* Control group: There is no health-related practice in the pensioners' club. No intervention will be made in the control group. After the experimental group's attempts are completed, a home visit is planned for the control group, and it is planned to make physical activity training, brochure, google fit application installation attempts.

ELIGIBILITY:
Inclusion Criteria:

* Independent elderly (Barthel activities of daily living index being above 60 points)
* Standardized Mini Mental Test Score above 24
* Not exercising regularly 3 days a week
* Not having a walking restriction by the physician
* To be at least primary school graduate
* Having a smart phone
* Having internet access at home or at work
* Ability to use the Internet

Exclusion Criteria:

* Dependent elderly people (Barthel activities of daily living index being below 60 points)
* Standardized Mini Mental Test Score below 24
* Exercising regularly 3 days a week
* Having a walking restriction by the physician
* Being illiterate
* Not having a smart phone
* Lack of internet access at home or at work
* Inability to use the Internet
* Diagnosis of heart failure

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Elderly health promotion scale | At the end of the 1st month.
  Elderly health promotion scale total score level
  * Health habits subdimension score level
  * Community participation subdimension score level
  * Health responsibility subdimension score level
  * Healthy eating subdimension score level
  * Regular exercise subdimension score level
  * Oral health subdimension score level All items in the scale are positive and have a four-point Likert scale (never (1), sometimes (2), often (3), always (4)). Scale scores range from 22 to 88, and it is stated that the higher the score, the more positive health promotion behaviors are shown.
Elderly health promotion scale | At the end of the 6st month.
  Elderly health promotion scale total score level
  * Health habits subdimension score level
  * Community participation subdimension score level
  * Health responsibility subdimension score level
  * Healthy eating subdimension score level
  * Regular exercise subdimension score level
  * Oral health subdimension score level All items in the scale are positive and have a four-point Likert scale (never (1), sometimes (2), often (3), always (4)). Scale scores range from 22 to 88, and it is stated that the higher the score, the more positive health promotion behaviors are shown.

SECONDARY OUTCOMES:
Physical Fitness and Exercise Activity Scale of Elderly Individuals Total score | At the end of the 1st month.
  The total score that can be obtained from the scale is min.34-max.136. Physical fitness subscale: 8-32 points. The higher the score obtained from the scale, the lower the physical fitness.
  Perceived obstacles subscale: 10-40 points. The lower the score, the higher the perceived obstacle is interpreted.
  Perceived motivators subscale: 8-32 points. The higher the scores, the lower the perceived motivators.
  Exercise frequency subscale: 7-28 points. Evaluation of the scale is as follows: "Strongly agree=1", "Agree= 2", "Disagree= 3", "Strongly disagree= 4". The evaluation of the exercise frequency subscale, which defines how often individuals participate in the defined activities, is "never / never =1", "once a week=2", "2-3 times a week =3", "every day =4".
Physical Fitness and Exercise Activity Scale of Elderly Individuals Total score | At the end of the 6st month.
  The total score that can be obtained from the scale is min.34-max.136. Physical fitness subscale: 8-32 points. The higher the score obtained from the scale, the lower the physical fitness.
  Perceived obstacles subscale: 10-40 points. The lower the score, the higher the perceived obstacle is interpreted.
  Perceived motivators subscale: 8-32 points. The higher the scores, the lower the perceived motivators.
  Exercise frequency subscale: 7-28 points. Evaluation of the scale is as follows: "Strongly agree=1", "Agree= 2", "Disagree= 3", "Strongly disagree= 4". The evaluation of the exercise frequency subscale, which defines how often individuals participate in the defined activities, is "never / never =1", "once a week=2", "2-3 times a week =3", "every day =4".

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK CİNGİL, Principal Investigator — https://erbakan.edu.tr/hemsirelikfak
Locations (1):
- Melikşah Retirees Club, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No